CLINICAL TRIAL: NCT00065650
Title: Pilot Study of Vedic Medicine for Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001324-01 (NIH)
Record Dates: First submitted 2003-07-30; First posted 2003-07-31 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; Vedic medicine; Ayurveda; Transcendental Meditation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Vedic Medicine
Behavioral: Vedic Medicine

SUMMARY:
The purpose of this study is to determine the feasibility and effectiveness of a multimodality Vedic Medicine treatment protocol for the management of newly diagnosed type 2 diabetes.

DETAILED DESCRIPTION:
Maharishi Vedic Medicine (MVM) represents a synthesis of Vedic sciences, including Ayur-Veda, into a single, comprehensive, natural approach to health care. The objectives of this phase II pilot trial are to determine the feasibility, acceptability, and safety of implementing a multi-modality MVM intervention for newly diagnosed type 2 diabetics, and to measure the impact of such a protocol on overall glycemic control.

ELIGIBILITY:
Inclusion criteria:

* Kaiser Permanente members
* Newly diagnosed type 2 Diabetes
* Baseline glycosylated hemoglobin level of 6.0-7.9.

Exclusion criteria:

* Pregnancy or nursing mother
* Currently taking warfarin
* Diagnosis of psychotic disorder or recent hospitalization for depression
* Unable to comply with or attend treatment sessions

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-07; Study Completion 2004-01

PRIMARY OUTCOMES:
HbA1C | 3 months

SECONDARY OUTCOMES:
Fasting Glucose | 3 and 6 months
Lipids | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Background] Elder C. Application of the cooperative health care clinic model for the delivery of complementary/ alternative care. The Permanente Journal. Winter 2003; 7(1):55-60.
- [Background] Elder C. Complementary and Alternative Medicine Symposium: Integrating CAM into clinical practice: The KP northwest story. The Permanente Journal, Fall 2002, 6(4):57-59
- [Result] Elder C, Aickin M, Bauer V, Cairns J, Vuckovic N. Randomized trial of a whole-system ayurvedic protocol for type 2 diabetes. Altern Ther Health Med. 2006 Sep-Oct;12(5):24-30. PMID 17017752
- See also: Kaiser Permanente Center for Health Research External Site — http://www.kpchr.org/public/default.asp